CLINICAL TRIAL: NCT05806125
Title: Clinical Value of the Fertility-preserving Surgery in Cervical Cancer -- the Feasibility of the 'Cuff-sleeve' Suture Method in the Ascending Branch of Uterine Artery Preserved Radical Trachelectomy
Brief Title: Clinical Value of the Fertility-preserving Surgery in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lu Huaiwu, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2022-038-01
Record Dates: First submitted 2023-03-19; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer
Keywords: computed tomography angiography; diameter of the supplying artery; fertility outcome; uterine blood supply pattern
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the postoperative group: All patients in the postoperative group will undergo computed tomography angiography (CTA) to evaluate the status of the preserved ascending branch and the residual uterine blood supply pattern after surgery.
- the preoperative group: Patients in the preoperative group will undergo CTA before RT to determine the uterine blood supply pattern in healthy individuals.

SUMMARY:
Purpose: To evaluate the clinical value of preserving the ascending branch of the uterine artery in improving the uterine blood supply after radical trachelectomy (RT). Method: This study will include 100 patients with early-stage cervical cancer, who undergo RT with the preservation of the ascending branch of the uterine artery. A new skill called the "cuff-sleeve" suture method is introduced to wrap the vagina around the stump cervix, wherein they are sutured using a 2-0 absorbable suture by placing two cross-stitches in the anterior and posterior wall, respectively, without piercing the cervical mucosa layer or damaging the uterine arteries. Study groups: The patients will be categorized into two groups. Patients in the postoperative group will undergo computed tomography angiography (CTA) after surgery and patients in the preoperative group will undergo CTA before RT. Data collection: Data regarding individual patient characteristics, International Federation of Gynecology and Obstetrics (FIGO) stage, histologic subtype, lymphovascular space involvement (LVSI) status, recurrence, CTA data, fertility results, and obstetric outcomes will be collected for the patients in the postoperative group. The CTA findings of the preoperative group will be obtained. Statistical methods: Statistical analyses were performed using IBM SPSS Statistics, version 26. The t-test is used for analyzing the continuous variables and the chi-squared test for categorical variables.

DETAILED DESCRIPTION:
Purpose: To evaluate the clinical value of preserving the ascending branch of the uterine artery in improving the uterine blood supply after radical trachelectomy (RT). Method: This study will include 100 patients with early-stage cervical cancer, who undergo RT with the preservation of the ascending branch of the uterine artery, at Sun Yat-sen Memorial Hospital, Sun Yat-sen University. The investigators attribute the uterine artery occlusion to the inevitable injury of the remaining uterine arteries during the ligation of the descending branch of the uterine artery and continuous or intermittent suturing. Hence, the investigators will carefully skeletonize the three branches of the uterine artery, ligates the vaginal and cervical branches, and preserves the ascending branch of the uterine artery under direct vision. Furthermore, a new skill called the "cuff-sleeve" suture method is introduced to wrap the vagina around the stump cervix, wherein they are sutured using a 2-0 absorbable suture by placing two cross-stitches in the anterior and posterior wall, respectively, without piercing the cervical mucosa layer or damaging the uterine arteries. Study groups: The patients will be categorized into two groups. All patients in the postoperative group will undergo computed tomography angiography (CTA) to evaluate the status of the preserved ascending branch and the residual uterine blood supply pattern after surgery. Patients in the preoperative group will undergo CTA before RT to determine the uterine blood supply pattern in healthy individuals. Data collection: Data regarding individual patient characteristics, International Federation of Gynecology and Obstetrics (FIGO) stage, histologic subtype, lymphovascular space involvement (LVSI) status, recurrence, CTA data, fertility results, and obstetric outcomes will be collected for the patients in the postoperative group. The CTA findings of the preoperative group will be obtained. The CTA data are mainly analyzed to determine the arteries supplying the uterus. The investigators consider a vessel as a supplying artery only when it is continuous from its origin up to the entry into the uterus and then branches. The uterine blood supply in patients is divided into three patterns based on the supplying vessels. The first is the ovarian artery-supplying pattern, wherein the residual uterus is supplied only by the ovarian arteries. The second is the hybrid-supplying pattern, in which an ovarian artery or a newly formed artery supplied the residual uterus along with the contralateral uterine artery. The third is the uterine artery-supplying pattern, wherein the residual uterus is supplied only by the uterine arteries. Furthermore, the diameter of the visualized supplying vessels is recorded. The diameters of the uterine and newly formed arteries are measured 2 cm before they enter the corpus uteri. However, the ovarian artery diameter is measured at its origin from the aorta ventralis, beside the external iliac artery, and 2 cm before it enters the corpus uteri since the ovarian arteries are convoluted. Statistical methods: Statistical analyses were performed using IBM SPSS Statistics, version 26. The t-test is used for analyzing the continuous variables and the chi-squared test for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female, ≥20 years old; 2. Clinical diagnosis of cervical cancer; 3. Received radical trachelectomy; 4. Have good compliance, and can complete the enrollment by the requirements of the trial; 5. Sign informed consent and agree to the collection and use of their data.

Exclusion Criteria:

* 1. Have received other anti-tumor treatments or received tumor surgery before enrollment; 2. With other malignant tumors; 3. With uncontrollable neurological, psychiatric, or mental disorders.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include 100 patients with early-stage cervical cancer, who undergo RT with the preservation of the ascending branch of the uterine artery. A new skill called the "cuff-sleeve" suture method is introduced to wrap the vagina around the stump cervix, wherein they are sutured using a 2-0 absorbable suture by placing two cross-stitches in the anterior and posterior wall, respectively, without piercing the cervical mucosa layer or damaging the uterine arteries.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The pattern of the uterine blood supply | The postoperative group will undergo CTA 3 months after surgery while the preoperative group will undergo CTA 1 week before the surgery.
  The first is the ovarian artery-supplying pattern, wherein the residual uterus is supplied only by the ovarian arteries. The second is the hybrid-supplying pattern, in which an ovarian artery or a newly formed artery supplied the residual uterus along with the contralateral uterine artery. The third is the uterine artery-supplying pattern, wherein the residual uterus is supplied only by the uterine arteries.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arbyn M, Weiderpass E, Bruni L, de Sanjose S, Saraiya M, Ferlay J, Bray F. Estimates of incidence and mortality of cervical cancer in 2018: a worldwide analysis. Lancet Glob Health. 2020 Feb;8(2):e191-e203. doi: 10.1016/S2214-109X(19)30482-6. Epub 2019 Dec 4. PMID 31812369
- [Background] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Clark R, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Huh WK, Lurain JR, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Cervical Cancer, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jan;17(1):64-84. doi: 10.6004/jnccn.2019.0001. PMID 30659131
- [Background] Dargent D, Martin X, Sacchetoni A, Mathevet P. Laparoscopic vaginal radical trachelectomy: a treatment to preserve the fertility of cervical carcinoma patients. Cancer. 2000 Apr 15;88(8):1877-82. PMID 10760765
- [Background] Cao DY, Yang JX, Wu XH, Chen YL, Li L, Liu KJ, Cui MH, Xie X, Wu YM, Kong BH, Zhu GH, Xiang Y, Lang JH, Shen K; China Gynecologic Oncology Group. Comparisons of vaginal and abdominal radical trachelectomy for early-stage cervical cancer: preliminary results of a multi-center research in China. Br J Cancer. 2013 Nov 26;109(11):2778-82. doi: 10.1038/bjc.2013.656. Epub 2013 Oct 29. PMID 24169350
- [Background] Bentivegna E, Maulard A, Pautier P, Chargari C, Gouy S, Morice P. Fertility results and pregnancy outcomes after conservative treatment of cervical cancer: a systematic review of the literature. Fertil Steril. 2016 Oct;106(5):1195-1211.e5. doi: 10.1016/j.fertnstert.2016.06.032. Epub 2016 Jul 16. PMID 27430207
- [Background] Querleu D, Morrow CP. Classification of radical hysterectomy. Lancet Oncol. 2008 Mar;9(3):297-303. doi: 10.1016/S1470-2045(08)70074-3. PMID 18308255